CLINICAL TRIAL: NCT06420960
Title: Rentabilité Diagnostique Des Montres connectées Par Rapport au Holter ECG Externe Dans l'Expertise Des Palpitations Fugaces Symptomatiques Sans Documentation électrocardiographique Per Critique.
Brief Title: Diagnostic Efficacy of Connected WAtch ECG Versus External Holter ECG
Acronym: WAHOE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: L'hôpital Nord-Ouest - Villefranche Villefranche sur Saône (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HNO23_0001; 2023-A01853-42 (Other: ANSM)
Record Dates: First submitted 2024-05-15; First posted 2024-05-20 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Heart Disease
Keywords: palpitations; yield diagnostic; connected watch; device; HOLTER ECG; monitoring; profitability
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- connected watch (Experimental): All patients will be equipped by HOLTER for 48-hour monitoring, with an event form to be filled in, at the same time as receiving a connected watch for a 6 -months period. They will be asked to record an ECG with the watch only when they experience symptoms that have included them in the study
  Interventions: Device: Wearing the connected watch
- HOLTER ECG 48 hours (Active Comparator): All patients will be equipped by HOLTER for 48-hour monitoring, with an event form to be filled in, at the same time as receiving a connected watch for a 6 -months period. They will be asked to record an ECG with the watch only when they experience symptoms that have included them in the study
  Interventions: Device: Wearing the connected watch

INTERVENTIONS:
Device: Wearing the connected watch — All patients will receive a connected watch from the research associate, along with instructions on its usage and support for creating an account on the Healtmate application using an anonymized e-mail address.
  They will be able to transmit up to 3 ECG tracings deemed to be per-critical. A follow-up phone call at 2- months will assess understanding of the device and its proper use, as well as the occurrence of adverse events and compliance.

SUMMARY:
Palpitations are a frequent reason for consultation (16% of total volume) and management in the emergency department.

Conventional diagnostic management in our establishment is based on a 48-hour external ECG holter, combined with a stress test if symptoms are triggered by physical activity.

The diagnostic difficulty lies in the frequency and duration of this transient symptom. At the time of consultation, the patient is often asymptomatic. The initial strategy is to demonstrate an electrocardiographic trace during the attack, in order to adapt management to the chosen etiology.

The HOLTER ECG is the gold standard, but it is not very cost-effective due to the infrequent and random nature of the onset of symptoms.

The advent of accessible connected tools such as connected watches seems to be an interesting alternative for acquiring a per-critical trace of symptoms. They are widely adopted by the general population, with ease of use by the individual and long monitoring times.

The main aim of the study is to establish the diagnostic cost-effectiveness of one or other of the two diagnostic strategies (rate of identification of the causal arrhythmia) at 6 months from the cardiological consultation.

ELIGIBILITY:
Inclusion Criteria:

* Any patient consulting for the main reason of palpitations; without a previous diagnosis of arrhythmia, unless the current symptomatology appears different from that associated with the previous rythmological diagnosis;
* Palpitations requiring cardiological consultation or emergency hospital treatment;
* Absence of suggestive diagnosis on intercritical 12-lead ECG (pre-excitation, AVB M2/3, high-grade atrioventricular block, non-sustained tachyventricular, atrial fibrillation with heart rate; 110 per minute, atrial tachycardia or flutter);
* Non-contributory stress test (no electrical abnormality, occurrence of arrhythmia or reproduction of palpitations) if isymptoms occur during exercise;
* Accepts to wear the watch all the time outside the charging time;
* Using a personal smartphone or tablet compatible with the Health Mate application and with an Internet connection;
* Affiliated with a social security system ;
* Providing dated and signed an informed consent form.

Exclusion Criteria:

* Refusal to wear the connected watch;
* Refusal to use the watch provided for the study because they use a personal connected watch;
* Unable to use the connected watch (lack of understanding of its use and rationale);
* No smartphone;
* Wearer of an implantable device (PM, ICD);
* Already known and treated arrhythmia with identical symptoms;
* Heart disease with indication for primary/secondary prevention implantable device;
* Associated syncope;
* Obvious extra-cardiac cause;
* Pregnant or breast-feeding woman;
* Inability to undergo study follow-up for geographical, linguistic, social or psychological reasons;
* Participating in another clinical study which can interfere with this study
* Patient under guardianship or deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2027-01-18 (Estimated); Study Completion 2027-02-17 (Estimated)

PRIMARY OUTCOMES:
Rate of diagnostic profitability of the connected watch compared with the conventional procedure (48-hour ECG Holter). | at 6 months or when the watch is returned, whether a diagnosis has been made or whether there have been 3 ECG transmissions that did not reveal any cardiac arrhythmia.
  The investigators will compare the diagnostic performance of the connected watch with the HOLTER ECG, by identifying a symptomatic arrhythmia, , in the purpose of a faster and adapted cardiological management.

SECONDARY OUTCOMES:
Type of diagnosis recorded. | at 6 months or when the watch is returned if a diagnosis has been made.
  A diagnosis is defined by the documentation of an objective cardiac arrhythmia (focal atrial tachycardia/atrial fibrillation HR >110 bpm/atrial fibrillation HR<110 bpm/atrial flutter/junctional tachycardia/sustained or non-sustained ventricular tachycardia/peak tachycardia/sinus tachycardia/ventricular fibrillation/high-degree conduction disorder) concomitant with the symptomatology motivating the initial consultation.
Rate of concomitant diagnoses with either device | at 6 months or when the watch is returned if a diagnosis has been made.
  Symptomatic objective cardiac arrythmia recorded with the smarwatch, the HOLTER or the both
Rate of causal non-rhythmological diagnosis (symptoms without pathological per-critical ECG tracing) | at 6 months or when the watch is returned if a diagnosis has been made or if there have been 3 ECG transmissions that did not reveal any cardiac arrhythmia.
  Rate of ECGs failing to explain symptomatology (no ECG abnormality detected ECG) Time Frame : at 6 months or when the watch is returned if a diagnosis has been made or if there have been 3 ECG transmissions that did not reveal any cardiac arrhythmia.
Medical/paramedical time per diagnosis and per patient | at 6 months or when the watch is returned, whether a diagnosis has been made or whether there have been 3 ECG transmissions that did not reveal any cardiac arrhythmia.
  Fitting of holter ECG equipment, handover of watch and explanation of how it works, analysis of holter/ ECG tracings, reconsultation)

CONTACTS AND LOCATIONS:
Locations (1):
- Hopitaux Nord-Ouest Villefranche Sur Saone, Gleizé, France

IPD SHARING:
Plan to Share IPD: Undecided
Confidentialité et protection de la vie privée : Le partage des données IPD pourrait compromettre la confidentialité et la protection de la vie privée des participants. Les données individuelles, même anonymisées, pourraient potentiellement être utilisées pour identifier des individus, en particulier dans le cas de petites cohortes ou de données sensibles.
  Sensibilité des données : Les données IPD inclusent des informations sensibles sur la santé. Le partage de telles données est soumis à des réglementations strictes sur la protection des données et nécessite des mesures supplémentaires pour garantir la sécurité et la confidentialité.
  Ressources et coûts : Le partage des IPD nécessite des ressources supplémentaires pour l'anonymisation, la gestion et la mise à disposition des données. Nous n'avons pas les ressources nécessaires pour effectuer ces tâches car notre budget est limité.